CLINICAL TRIAL: NCT03951480
Title: Care of AcromioClavicular Arthropathy in Manual Medicine Versus Corticosteroid Infiltration : Non-inferiority Study
Brief Title: Care of AcromioClavicular Arthropathy in Manual Medicine Versus Corticosteroid Infiltration (ACAM)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion target not met. Inclusion period not extended.
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHD 023-19
Record Dates: First submitted 2019-04-25; First posted 2019-05-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Acromioclavicular Arthropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual medicine (Experimental)
  Interventions: Other: Manual medicine
- Corticosteroids infiltration (Active Comparator)
  Interventions: Drug: Corticosteroids infiltration

INTERVENTIONS:
Other: Manual medicine — At a rate of 3 sessions of a maximum of 30 minutes each at one week interval. Depending on the clinical evolution, it is possible to stop manual medicine sessions according to the therapist's assessment as in current practice. If the patient has an EVA pain of activity < 2, manipulations will not be continued. The patient being considered as not very symptomatic.
  Arms: Manual medicine
Drug: Corticosteroids infiltration — A unique echo-guided infiltration of one syringe of 1 mL of cortisone product
  Arms: Corticosteroids infiltration

SUMMARY:
Acromioclavicular pains are one of the etiologies of shoulder pains, the prevalence of which is relatively high, ranging from 5 to 47% in the general population. The cause is usually degenerative, occurring mainly after the age of 40, especially in male manual workers. This pathology is described as the great forger of the shoulder, ignored by clinicians because it is often uninvestigated, whereas an interrogation and a complete clinical examination are sufficient to make the diagnosis.

Acromioclavicular pathologies are better known to orthopaedic surgeons, particularly in traumatic pathologies but also in degenerative pathologies. However, before operating on acromioclavicular osteoarthritis, interventions whose results are sometimes disappointing, a well-managed medical treatment usually helps to relieve pain.

The precise clinical examination and a radiological examination focused on the joint make it possible to diagnose acromioclavicular arthropathy, the key is to think about it and look for it.

Care includes explanation of the diagnosis, drug treatments, physiotherapy techniques and self-exercise as well as osteoarticular manipulations, which are less frequently practiced or performed in isolation outside the medical setting.

The results of the different treatments have been little studied, with studies that don't always allow us to distinguish several etiologies of shoulder pains. Most studies compare surgical techniques with each or with medical techniques. However, there are very few studies comparing traditional medical care with manual medicine.

In order to compare the different non-surgical therapies for the care of acromioclavicular arthropathies of degenerative origin, the investigators propose a dedicated study.

This is a non-inferiority, prospective, open, randomized, two-armed study comparing the efficacy of manipulations by a physician with a training in manual medicine versus cortisone infiltration Under ultrasound control.

After diagnosis of degenerative pathology of the acromioclavicular joint, patients meeting the inclusion criteria will be randomized to the infiltration arm or to the manipulations arm.

The assessment will be based on the pain during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30 to 80 years old
* Shoulder ou proximal arm pain with elective pain on palpation of the acromioclavicular joint + Positive cross arm test + Positive O'Brien test
* NEER test negative: pain < 4
* Symptomatic acromioclavicular arthropathy confirmed on radiography
* Pain at rest or activity (EVA ≥ 4) for more than 3 months
* Patient with the ability to understand the protocol and who has signed an informed consent
* Patient with social security coverage

NSAID or per os or topical analgesics may also be taken at the same time as participation in the study.

Exclusion Criteria:

* Contraindication to scapular or cervical manipulation
* Contraindication to infiltration (unbalanced diabetes, unbalanced hypertension, ongoing infections)
* Local or generalized infection
* Known history of severe bleeding disorders, anticoagulant therapy in progress (AVK, NACO) and Plavix
* Severe hypertension > 160/100 mmHg and/or uncontrolled
* Unbalanced diabetes (last HbA1c > 8,5%)
* Live vaccines in the 3 months preceding the study and throughout the study (MMR, yellow fever, Bacillus Calmette-Guerin, oral polio vaccine)
* Known hypersensitivity to Diprosten® including its excipients (methyl parahydroxybenzoate, propylparahydroxybenzoate, benzyl alcohol)
* Inflammatory rheumatism (RA, PPR, SPA)
* Microcrystalline rheumatism of the shoulder (drop ou CCA)
* History of surgery or trauma that justified surgical or arthroscopic intervention of the shoulder
* Previous infiltrations of the shoulder less than 6 months old
* Patient with a diagnosis of associated fibromyalgia
* Severe cases of water retention and/or sodium (hypernatremia), particularly in cases of heart failure, decompensated liver failure (edema, ascites) and severe renal failure
* Immunocompromised or hemodialysed patients
* Pregnant or breastfeeding women
* Patient with reproductive capacity and refusing effective contraception
* Patients Under guardianship, curators, or deprived of liberty
* Patients participating in another interventional clinical research protocol involving a drug or medical device
* Patients unable to follow the protocol, as determined by the investigator's judgment

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
The main objective of this study is to compare the medium-term efficacy on pain of manual medical care of degenerative acromioclavicular arthropathy versus infiltrative care Under ultrasound detection with a cortisone product | At three months
  Use of a visual analogue scale to measure pain

CONTACTS AND LOCATIONS:
Overall Officials: Alexia MICHAUT, Principal Investigator — CHD Vendée
Locations (1):
- Centre Hospitalier Départemental Vendée, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michaut A, Planche L, Auzanneau L, Cormier G. Management of acromioclavicular joint disease by manual therapy versus corticosteroid injections: the protocol of a non-inferiority study. BMJ Open. 2020 Dec 10;10(12):e034439. doi: 10.1136/bmjopen-2019-034439. PMID 33303428